CLINICAL TRIAL: NCT05560854
Title: A Feasibility Study of Internet Delivered Prolonged Exposure for Patients Wit Post-traumatic Stress Disorder
Brief Title: A Feasibility Study of Internet Delivered Prolonged Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Maria Bragesjo, Principal investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-03465-01
Record Dates: First submitted 2022-09-23; First posted 2022-09-29 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Prolonged exposure; Internet-delivered; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Prolonged exposure will be offered in a digital format with therapist support for ten weeks. Treatment comprises of psychoeducation, rationales, in vivo exposure, imaginal exposure, problems that can arise during exposure, hot spots and relapse prevention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet delivered prolonged exposure (Experimental): Internet delivered prolonged exposure for ten weeks with therapist support.
  Interventions: Behavioral: Internet delivered prolonged exposure

INTERVENTIONS:
Behavioral: Internet delivered prolonged exposure — Internet delivered prolonged exposure for ten weeks with therapist support.

SUMMARY:
The primary objective with this study is to investigate the feasibility and acceptability of ten weeks of internet delivered prolonged exposure delivered through a digital platform with therapist support. The secondary objective is to investigate preliminary effects of internet delivered prolonged exposure in terms of reducing symptoms of post-traumatic stress, depression and increase quality of life.

DETAILED DESCRIPTION:
The investigators will investigate internet delivered prolonged exposure delivered as a ten-week treatment comprising of six modules (psychoeducation/rational, in vivo exposure, imaginal exposure, common problems during exposure, hot spots and relapse prevention). The feasibility and acceptability and preliminary effects of treatment- and assessment procedures will be evaluated using a within-group design with repeated measurements and qualitative interviews. Recruitment is designed to be broadly inclusive with minimal exclusion criteria. Patients will be recruited from a psychiatric clinic specialized in PTSD in Stockholm, Sweden and by advertisements in newspapers and social media.

ELIGIBILITY:
Inclusion Criteria:

* Currently primary diagnosis PTSD according to DSM-5 diagnostic criteria for PTSD
* ≥ 18 years
* Fluent in Swedish
* Signed informed consent

Exclusion Criteria:

* PTSD is not the primary concern
* Initiation or adjustment of any psychotropic medication within the last 4 weeks prior to commencement of treatment
* Ongoing substance dependence
* Current suicide risk meriting crisis intervention
* Psychotic disorder
* Ongoing trauma-focused psychological treatment
* Ongoing trauma-related threat (e.g. living with a violent spouse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-09-09 (Actual); Study Completion 2023-09-09 (Actual)

PRIMARY OUTCOMES:
Number of imaginal exposures made by the participant during the treatment period | Through the treatment period, up to 10 weeks
  Number of imaginal exposures made by the participant during the treatment
Number of in vivo exposures made by the participant during the treatment period | Through the treatment period, up to 10 weeks
  Number of in vivo exposures made by the participant during the treatment period
The proportion of participants that conducts the weekly measures and further assessment points | Through study completion up to the 6 months follow up]
  The proportion of participants that conducts the weekly measures and further assessment points
The proportion of participants that go through the entire treatment period | Completion of the treatment period, ten weeks
  The proportion of participants that go through the entire treatment period
Adverse events related to the treatment | Through study completion, up to the 6 months follow up
  Treatment acceptability
Number of drop-outs from treatment | Completion of the treatment period, up to 10 weeks
  Treatment acceptability
Participants experience/satisfaction with treatment and assessment procedures through qualitative interviews | Completion of the treatment period up to the 6-month follow up
  Qualitative interviews
Participants satisfaction with treatment, assessed by The Client Satisfaction Questionnaire (CSQ-8). | Completion of the treatment period, up to 10 weeks
  The CSQ-8 yields a single score measuring a single dimension of overall satisfaction. An "overall score" is calculated by summing the score on each of the eight scale item. Scores range from 8 to 32, with higher values indicating higher satisfaction.

SECONDARY OUTCOMES:
Change in PTSD symptoms as assessed by the Clinician Administered PTSD Scale (CAPS-5) | Baseline, 1 month and 6 months follow up
  The CAPS-5 is structured interview that assesses the Diagnostic and Statistical Manual of Mental Disorders version 5 (DSM-5) criteria for PTSD (Weathers et al., 2013). Each item is rated on a severity scale ranging from 0 (Absent) to 4 (Extreme/incapacitating) and combines information about frequency and intensity for each of the 20 symptoms. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.
Change in PTSD symptoms as assessed by the PTSD Check List - DSM-5 (PCL-5) | Baseline, weekly through 10 weeks of treatment, post-treatment (immediately after treatment completion at 10 weeks), and the 1 month and 6 months follow up.
  The PCL-5 is a 20-item self-report measure based upon the Diagnostic and Statistical Manual (DSM-5) criteria for PTSD. Total Score (Range 0-80 with higher scores representing more PTSD symptoms.
Change in ICD-11 PTSD and complex PTSD symptoms as assessed by the International Trauma Questionnaire (ITQ). | Baseline, weekly through 10 weeks of treatment, post-treatment (immediately after treatment completion at 10 weeks), and the 1 month and 6 months follow up.
  The ITQ includes six items measuring each PTSD symptom cluster and these items measure how bothersome each symptom has been in the past month. The ITQ also includes six items measuring each 'Disturbance in Self- Organization' (DSO) symptom in complex PTSD. These items measure how a respondent typically feels, thinks about oneself, and relates to others. The PTSD and DSO symptoms are accompanied by three items measuring associated functional impairments in the domains of social, occupation, and other important areas of life. All items are answered on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Extremely). Thus, PTSD and DSO symptom scores range from 0 to 24 and CPTSD symptom scores range from 0 to 48. Higher scores represents more PTSD and complex PTSD symptoms.
Change in depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline, post-treatment (immediately after treatment completion at 10 weeks), and the 1 month and 6 months follow up.
  The PHQ-9 is a widely used and well-validated instrument for measuring the severity of depressive symptoms. Scores are calculated based on how frequently a person experiences 9 symptoms of depression ranging from "not at all" response is scored as 0; "several days" response is 1; "more than half the days" response is 2; and "nearly every day" response is 3. Higher scores represents more depressive symptoms.
Change in quality of life measured by Euroqol, EQ-5D | Baseline, post-treatment (immediately after treatment completion at 10 weeks), and the 1 month and 6 months follow up.
  Change in overall health from baseline to post treatment and follow up . EQ-5D is a standardized self-report measure of overall health status measured in terms of five dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using a three-level scale: 1 having no problems, 2 having some problems and 3 having extreme problems. A higher score indicate worse severity.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Bragesjö, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Traumaprogrammet, Psykiatri Sydväst, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bragesjo M, Ivanov VZ, Andersson E, Ruck C. Exploring the feasibility and acceptance of huddinge online prolonged exposure therapy (HOPE) for severe and complex PTSD. Eur J Psychotraumatol. 2024;15(1):2320607. doi: 10.1080/20008066.2024.2320607. Epub 2024 Mar 4. PMID 38436944